CLINICAL TRIAL: NCT04536142
Title: Evaluation of Changes in Brain Connectivity After Tumor Resection
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: Great Plains IDeA-CTR (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0155-20-EP
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brain tumors: Subjects with operable supratentorial brain tumors
  Interventions: Diagnostic Test: MRI; Diagnostic Test: neuropsychological tests and qualitative assessment
- Healthy subjects: Healthy subjects
  Interventions: Diagnostic Test: MRI; Diagnostic Test: neuropsychological tests and qualitative assessment

INTERVENTIONS:
Diagnostic Test: MRI — A research MRI scan will be performed within 1 week prior to surgery and again 2 weeks after surgery. The surgical removal of the brain tumor(s) is not a component of this research. The MRI scan will perform both programs (diffusion MRI, resting state MRI) during the same single session. The healthy controls will obtain identical research scans with the second session between two and three weeks following the first session, since they will not undergo a surgery.
Diagnostic Test: neuropsychological tests and qualitative assessment — Neuropsych Tests: COWA, Trails, RCFT, RAVLT, WMS-III subtests, NAB Digits, Grooved Pegboard, Stroop Color Word Test, verbal and spatial working memory, WRAT-IV, Word Reading subtest.
  Standardized quality of life measures: MDASI-BT, FACT-Br, FrSBe

SUMMARY:
This study is being done to see the changes in structural and functional connectivity that happen in the brain of patients undergoing brain tumor surgery.

DETAILED DESCRIPTION:
The purpose of this study is to visualize and quantify changes in the brain of patients undergoing brain tumor surgery through high-quality, high-resolution structural and functional brain imaging and brain connectivity measures. To understand the effects of the primary treatment for brain tumors, the investigators will determine changes in brain connectivity after surgery and correlate this with neurologic status. The investigators will prospectively collect brain imaging (MRI) and clinical data in brain tumor patients before and after removal of their tumor. Any adult patient with a brain tumor (primary or metastatic) for whom surgery to remove the tumor is planned is eligible. The investigators plan for recruitment of 30 subjects. This will include 27 subjects with brain tumors and 3 healthy controls. Both clinical and imaging data will be collected for tumor and healthy subjects. A two-part research scan (diffusion MRI and resting state functional MRI) will be performed within 1 week prior to surgery and again 2 weeks after surgery. The healthy controls will obtain identical research scans with the second session two weeks following the first session. Subjects will be also administered Neurocognitive and Qualitative Assessments at two time intervals, pre- and post-surgery (2 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Brain tumor subjects (27)

   * informed consent
   * age equal to or greater than 19 years (age of majority in Nebraska)
   * brain tumor that requires surgery
   * primary or metastatic brain tumor
2. Healthy subjects (3)

   * informed consent
   * age equal to or greater than 19 years (age of majority in Nebraska)
   * healthy subject with no know neurocognitive deficiencies

Exclusion Criteria:

* any contraindication to MRI (i.e. implanted devices)
* inappropriate body habitus for MRI
* no capacity to understand the study the study or consent to it
* positive pregnancy test in females
* end stage renal disease or severe renal dysfunction
* severe anxiety disorder
* metabolic encephalopathy
* significant medical co-morbidities precluding a safe surgery
* need for sedation for MRI

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oncologists and neurosurgeons may identify their patients for potential inclusion as brain tumor subjects. The "word-of-mouth" approach will be used to identify potential healthy subjects for this study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Brain connectivity changes | MRI scan will be performed within 1 week prior to surgery and again 2 weeks after surgery.
  With both the functional and structural connectomes created, the investigators will compute graph network measures before and after surgical resection and assess both nodal and global network measures.
Neurocognitive changes | Cognitive tests will be performed within 1 week prior to surgery and again 2 weeks after surgery.
  Meyers Neuropsychological Battery: Published reliable change indices (RCI) will be used to control for practice effects between the assessment points for all Meyers Neuropsychological Battery (MNB) subtests.
  QOL inventories: Differences in scores at baseline, relative to treatment phase, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Aizenberg, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No